CLINICAL TRIAL: NCT06425133
Title: Impact of Regorafenib in Combination With Multimodal Metronomic Chemotherapy on Progression-free Survival Compared With Standard Regorafenib for the Treatment of Chemo-resistant Metastatic Colorectal Cancers
Brief Title: Regorafenib in Combination With Multimodal Metronomic Chemotherapy for Chemo-resistant Metastatic Colorectal Cancers
Acronym: CARE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Groupement Interrégional de Recherche Clinique et d'Innovation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/805
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Regorafenib; metronomic chemotherapy; colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Blood Specimen Collection; Biopsy; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regorafenib (Active Comparator): • Regorafenib will be administered 3 weeks out of 4 (1 cycle corresponding to 4 weeks) until progression or unacceptable toxicity.
  For the first cycle: Regorafenib will be administered according to the "REDOS" schedule week 1: 80 mg regorafenib daily week 2: 120 mg regorafenib daily week 3: 160 mg regorafenib daily week 4 : no regorafenib
  For the following cycles: regorafenib will be administered at 160mg in the absence of significant toxicity during cycle 1 or at a 80/120mg daily dose according to toxicity observed with the last dose used in the first cycle.
  Interventions: Procedure: Blood sample; Other: Quality of life questionnaires; Procedure: Biopsy; Drug: Regorafenib
- Regorafenib+ metronomic chemotherapy + aspirin (Experimental): • Regorafenib will be administered 3 weeks out of 4 (1 cycle corresponding to 4 weeks) until progression or unacceptable toxicity.
  For the first cycle: Regorafenib will be administered according to the "REDOS" schedule: week 1: 80 mg daily week 2: 120 mg daily week 3: 160 mg daily week 4 : OFF. For the following cycles: regorafenib will be administered at 160mg in the absence of significant toxicity during cycle 1 or at a 80/120mg daily dose according to toxicity observed with the last dose used in the first cycle.
  * Metronomic chemotherapy will be administrated as following:Cyclophosphamide: 50 mg per os, daily, for 6 months,Capecitabine: 625mg/m²/orally twice daily, for 6 months.
  * Low-dose Aspirin: 75 mg orally, daily, until progression.
  Interventions: Procedure: Blood sample; Other: Quality of life questionnaires; Procedure: Biopsy; Combination Product: Regorafenib + metronomic chemotherapy

INTERVENTIONS:
Procedure: Blood sample — Blood sample for plasma collection, Blood sample for ctDNA (circulating tumoral DNA) collection
Other: Quality of life questionnaires — EORTC QLQ-C30 questionnaire (Quality of life questionnaire Cancer 30) CR29 questionnaire (Colo-rectal cancer 29) EQ-5D5L questionnaire (EuroQol-5 Dimensions, 5 levels): repeated measures at baseline, M2, M4, M6, M8, M10, M12 and during the end of treatment visit and during the follow-up
Procedure: Biopsy — Fresh tumor biopsy at baseline and week 8
Drug: Regorafenib — For the first cycle: Regorafenib will be administered according to the "REDOS" schedule: week 1: 80 mg regorafenib daily week 2: 120 mg regorafenib daily week 3: 160 mg regorafenib daily week 4 : OFF. For the following cycles: regorafenib will be administered at 160mg in the absence of significant toxicity during cycle 1 or at a 80/120mg daily dose according to toxicity observed with the last dose used in the first cycle.
  Arms: Regorafenib
Combination Product: Regorafenib + metronomic chemotherapy — • Regorafenib will be administered 3 weeks out of 4 (1 cycle corresponding to 4 weeks) until progression or unacceptable toxicity.
  For the first cycle: Regorafenib will be administered according to the "REDOS" schedule: week 1: 80 mg regorafenib daily week 2: 120 mg regorafenib daily week 3: 160 mg regorafenib daily week 4 : OFF. For the following cycles: regorafenib will be administered at 160mg in the absence of significant toxicity during cycle 1 or at a 80/120mg daily dose according to toxicity observed with the last dose used in the first cycle.
  * Metronomic chemotherapy will be administrated as following:Cyclophosphamide: 50 mg per os, daily, for 6 months,Capecitabine: 625mg/m²/orally twice daily, for 6 months.
  * Low-dose Aspirin: 75 mg orally, daily, until progression.
  Arms: Regorafenib+ metronomic chemotherapy + aspirin

SUMMARY:
The main objective is to evaluate the impact of a Regorafenib combined with metronomic chemotherapy (capecitabine and cyclophosphamide) and low-dose aspirin compared to standard Regorafenib treatment in patients with metastatic colorectal cancer by assessing progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven metastatic colorectal cancer in progression after previous standard treatments (5FU, CPT11 (Irinotecan), oxaliplatin, anti-VEGF (vascular endothelial growth factor), trifluridine/tipiracil, anti-EGFR (epidermal growth factor receptor) therapy if KRAS (Kirsten rat sarcoma) and NRAS WT (wild type), anti-BRAF therapy if BRAF V600E mutated, and anti-PD1 (Programmed Death-1) if MSI-H (microsatellite instability) /dMMR (deficient MisMatch Repair) tumor, or not considered as candidate for these treatments.
2. Life expectancy of at least 3 months
3. Female or male with age >18 years old
4. Performance status = 0 or 1 (Annex 1)
5. Measurable disease defined according to RECIST v1.1 guidelines (scanner or MRI)
6. Adequate bone marrow, liver and renal functions.

   1. Haemoglobin ≥ 9 g/dL; absolute neutrophil count (ANC) ≥ 1.5 x 109/L; platelets ≥ 100 x 109/L
   2. Total serum bilirubin ≤ 1.5 times upper normal value (ULN), serum alkaline phosphatase < 5 times ULN, aminotransferases (AST/ALT) ≤ 3 × ULN in absence of hepatic metastasis or ≤ 5 if presence of hepatic lesions
   3. Cockcroft glomerular filtration rate > 50 ml/min
   4. Proteinuria <2+ (dipstick urinalysis) or ≤1g/24hour
7. No contraindication to Iodine contrast media injection during CT
8. For female patients of childbearing potential, negative pregnancy test within 14 days before starting the study drug. Men and women are required to use adequate birth control during the study (when applicable),
9. Signed and dated informed consent,
10. Ability to comply with the study protocol, in the Investigator's judgment.
11. Registration in a national health care system (CMU included).

Exclusion Criteria:

1. Diagnosis of additional malignancy within 2 years prior to the inclusion (exception of curatively treated basal cell carcinoma of the skin and/or curatively resected in situ cervical and/or bladder cancer),
2. Current participation in a study of an investigational agent or in the period of exclusion
3. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before inclusion in the trial ;
4. Patient under judicial protection (curators, autorship) and/or deprived of freedom,
5. Previous exposition to regorafenib or anti-angiogenic treatment other than bevacizumab and aflibercept
6. Treatment with any other investigational medicinal product within 28 days prior to study entry, EXCEPT for ASPIRIN,
7. Systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy, and hormonal therapy during this trial or within 3 weeks,
8. Chronic treatment with drug potentially interacting with regorafenib i.e. CYP3A4, CYP2C9 or UGT1A9 (UDP-glucuronosyltransferase 1-9) inductor/inhibitor; Epileptic disorder requiring medication; Recent or concomitant treatment with brivudine,
9. Complete deficit in dihydropyrimidine dehydrogenase (DPD),
10. Known hypersensitivity to any of the study drugs, study drug classes or excipient in the formulation:

    * History of severe and unexpected reactions to fluoropyrimidine therapy,
    * History of asthma induced by the administration of salicylates or substances with a similar action, notably non-steroidal anti-inflammatory medicines,
    * Mastocytosis, for whom the use of acetylsalicylic acid can cause severe hypersensitivity reactions,
11. Unresolved toxicity higher than CTCAE (v5) Grade 1 attributed to any prior therapy/procedure excluding alopecia, hypothyroidism and oxaliplatin induced neuropathy ≤ Grade 2,
12. Subject unable to swallow oral medications or any malabsorption condition,
13. Inadequate organ functions:

    * known cardiac failure of unstable coronaropathy, respiratory failure, or uncontrolled infection or another life-risk condition
    * Congestive Heart Failure ≥ New York Heart Association (NYHA) class 2,
    * Myocardial infarction less than 6 months before start of study drug, unstable angina (anginal symptoms at rest), new-onset angina (begun within the last 3 months), Cardiac arrhythmias requiring anti-arrhythmic therapy (beta-blockers or digoxin are permitted),
    * Uncontrolled hypertension (defined by systolic blood pressure ≥ 150 mmHg and/or diastolic pressure ≥ 100 mmHg despite optimal medical management), or history of hypertensive crisis, or hypertensive encephalopathy
    * Pleural effusion or ascites that causes respiratory compromise (≥ CTCAE grade 2 dyspnea),
    * Interstitial lung disease with ongoing signs or symptoms,
    * Ongoing infection >grade 2 CTCAE V5,
    * Dehydration CTCAE v5 grade ≥1,
    * Urinary tract obstruction
14. Constitutional or acquired hemorrhagic disease:

    * Any haemorrhage or bleeding event ≥ CTCAE Grade 3 within 4 weeks prior to the start of study medication,
    * History of abdominal fistula, GI perforation, intra-abdominal abscess or active GI bleeding within 6 months prior to inclusion,
    * Serious, Non-healing wound, active peptic ulcer or untreated bone fracture,
    * Major surgical procedure, open biopsy or significant traumatic injury within 28 days before start of study medication,
15. Planned surgical procedure within the first month of treatment or any procedure that might change the timing of regorafenib administration during the first month of treatment,
16. Known History of human immunodeficiency virus (HIV) infection; Active hepatitis B or C or chronic hepatitis B or C requiring treatment with antiviral therapy,
17. Receipt of yellow fever vaccine within 28 days prior to study,
18. History of organ allograft,
19. Pregnant or breast-feeding subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the impact of a Regorafenib combined with metronomic chemotherapy and low-dose aspirin compared to standard Regorafenib treatment by assessing progression-free survival | 5 months average
  Progression-free survival (PFS): defined as the time from the randomization to objective disease progression as per RECIST v1.1 or death from any cause, whichever occurs first. The time of the progression or recurrence event is determined using the first date when there is documented evidence that the criteria have been met, even in situations where progression is observed after one or more missed visits, treatment discontinuation, or new anti-cancer treatment.
  Patients with no defined events observed during the follow up period will be censored at the date of last news

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU d'Auxerre, Auxerre
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - CH de Colmar, Colmar
  - Centre Georges-François Leclerc (CGFL), Dijon
  - Hôpital Robert Schuman, Metz
  - Hôpital Nord Franche-Comté, Montbéliard
  - CHU de Montpellier, Montpellier
  - CHU de Reims - Hôpital Robert Debré, Reims
  - Clinique Privée de Strasbourg, Strasbourg
  - ICANS, Strasbourg